CLINICAL TRIAL: NCT02503020
Title: Effects of Different Arachidonic Acid Supplementation on Psychomotor Development in Very Preterm Infants, a Randomized Controlled Trial
Brief Title: Arachidonic Acid Supplementation in Very Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Health Research Institute of Santiago (Other)
Responsible Party: Principal Investigator, Ayham alshweki, Principal Investigator, Health Research Institute of Santiago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: Ayham
Record Dates: First submitted 2015-07-14; First posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Impaired Psychomotor Development
Keywords: Arachidonic acid; Omega-6/omega-3 ratio; Preterm infants nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Preterm infants formula A Pretarm infants were fed on formula with Arachidonic acid (0.6%) and Docosahexaenoic acid (0.3%)
  Interventions: Dietary Supplement: Preterm infants formula A
- Group B (Active Comparator): Preterm infants formula B Pretarm infants were fed on formula with Arachidonic acid (0.3%) and Docosahexaenoic acid (0.3%)
  Interventions: Dietary Supplement: Preterm infants formula B

INTERVENTIONS:
Dietary Supplement: Preterm infants formula A — Group A will receive a preterm infants formula supplemented with AA (0.6%) and DHA (0.3%) until they have three months corrected age. At 3 and 6 months of corrected age, we changed the type of milk according to the nutritional requirements, but maintained the same ratio of AA and DHA (2/1) until one year corrected age.
  Arms: Group A
Dietary Supplement: Preterm infants formula B — Group B will receive other Preterm infants formula very similar, but with AA (0.3%) and DHA (0.3%) also until they have three months corrected age.
  At 3 and 6 months of corrected age, we changed the type of milk according to the nutritional requirements, but maintained the same ratio of AA and DHA (1/1) until one year corrected age.
  Arms: Group B

SUMMARY:
Long-chain polyunsaturated fatty acids (LCPUFAs), arachidonic acid (AA omega-6; 20:4ω-6), and docosahexaenoic acid (DHA omega-3; 22:6ω-3), are required for the formation of non-myelinated cell membranes in the central nervous system, including in the retina, hence the great importance of them for appropriate visual and cognitive development.

In this study, the investigators assessed anthropometric, visual, auditory, and psychomotor development in very preterm infants who had diets supplemented with different LCPUFA amount of AA to support the importance of sufficient AA values in formula.

DETAILED DESCRIPTION:
the investigators carried out a prospective randomized controlled double blinded trial in order to study nutritional supplements for preterm infants <1500 grams and/or <32 weeks gestational age (GA) who were born in clinical University Hospital of Santiago de Compostela (CHUS). They were enrolled for a period of 14 months (from July 2011 to August 2012) and followed up from birth until 2 years of age. Milk formulas were provided either as adjunct to insufficient amount of breast milk, or as full formula feeding. Breastfeeding was actively encouraged. Patients were randomized into one of the two formula groups, depending on the type of formula they were to receive. Group A's formula was supplemented with DHA (0.3% of all fatty acids) and AA (0.6%) with an ω-6/ω-3 ratio of 2/1. Group B's formula was supplemented with DHA (0.3%) and AA (0.3%) with an ω-6/ω-3 ratio of 1/1.

Primary outcome:

Assessment of psychomotor development with the Brunet Lézine scale at 2 years of age (Early Care Unit CHUS)

Secondary outcomes:

Physical examination and anthropometric measurements (weight, length, and head circumference) at birth and at 3, 6, 9, 12, 18, and 24 months of age (Neonatology Unit CHUS) Blood levels of fatty acids in the first week of life and at 3 months, 6 months, and 12 months. (Metabolic Unit. Hospital de Cruces, Bilbao) Visual- and auditory-evoked potentials at 6 and 12 months of age (Neurophysiology Unit CHUS)

ELIGIBILITY:
Inclusion Criteria:

* Living infants who were less than 1500 grams and/or less than 32 weeks gestational age, and whose parents accepted and subscribed the informed consent

Exclusion Criteria:

* Preterm infants with any severe malformation.
* Extremely preterm infants with a gestational age of less than 25 weeks.
* Infants whose parents could not complete the follow-up process in our study center.
* Preterm infants with severe intraventricular hemorrhage or periventricular leukomalacia (more than grade 2).
* Neonates who did not need supplementary milk nutrition, i.e. breastfed-only children.

Ages: 1 Minute to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Psychomotor development | From september 2013 to november 2014 (at two years of corrected age)
  Evaluation of psychomotor development by making Brunet-Lezine scale at 2 years of corrected age.

SECONDARY OUTCOMES:
Levels of fatty acids in plasma | From october 2011 to november 2013 (from 3 months to 1 years old)
  Blood samples were obtained from study children to study the levels of fatty acids in plasma at 3 , 6 and 12 months of life
Visual- and auditory-evoked potentials | From january 2012 to February 2013 (from 6 months to 1 years old)
  Visual- and auditory-evoked potentials were studied with special scale at 6 and 12 months of life
Weight | From october 2011 to november 2014 (from 6 months to 2 years old)
  Weight at 3, 6, 9, 12, 18, and 24 months of life
Length | From october 2011 to november 2014 (from 6 months to 2 years old)
  Length at 3, 6, 9, 12, 18, and 24 months of life
Head circumference | From october 2011 to november 2014 (from 6 months to 2 years old)
  Head circumference at 3, 6, 9, 12, 18, and 24 months of life

REFERENCES:
- [Derived] Alshweki A, Munuzuri AP, Bana AM, de Castro MJ, Andrade F, Aldamiz-Echevarria L, de Pipaon MS, Fraga JM, Couce ML. Effects of different arachidonic acid supplementation on psychomotor development in very preterm infants; a randomized controlled trial. Nutr J. 2015 Sep 30;14:101. doi: 10.1186/s12937-015-0091-3. PMID 26424477